CLINICAL TRIAL: NCT01775579
Title: Randomized, Open Label, Multiple-Dose, 6-sequence, 3-period, Crossover Study to Evaluate a Pharmacokinetic Drug Interaction Between Metformin Hydrochloride and Rosuvastatin Calcium in Healthy Male Subjects
Brief Title: Evaluating a Pharmacokinetic Drug Interaction Between Metformin Hydrochloride and Rosuvastatin Calcium
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hanmi Pharmaceutical Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HM-MERO-101
Record Dates: First submitted 2013-01-23; First posted 2013-01-25 (Estimated); Last update posted 2013-08-23 (Estimated); Status verified 2013-08

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus | interventions — Rosuvastatin Calcium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Crestor tablet 20 mg (Experimental): Crestor tablet 20 mg single--->wash out---->Glucophage SR tablet 750 mg single---->washout--->Glucophage SR tablet 750 mg, Crestor tablet 20 mg both
  Interventions: Drug: Glucophage SR tablet 750 mg, Crestor tablet 20 mg
- Glucophage SR tablet 750 mg and Crestor tablet 20 mg both (Experimental): Glucophage SR tablet 750 mg, Crestor tablet 20 mg both--->wash out---->Glucophage SR tablet 750 mg single------>washout--->Crestor tablet 20 mg single
  Interventions: Drug: Glucophage SR tablet 750 mg, Crestor tablet 20 mg
- Glucophage SR tablet 750 mg (Experimental): Glucophage SR tablet 750 mg single --->wash out---->Crestor tablet 20 mg single---->washout--->Glucophage SR tablet 750 mg, Crestor tablet 20 mg both
  Interventions: Drug: Glucophage SR tablet 750 mg, Crestor tablet 20 mg

INTERVENTIONS:
Drug: Glucophage SR tablet 750 mg, Crestor tablet 20 mg

SUMMARY:
We investigate the potential pharmacokinetic drug-drug interaction between metformin extended release and rosuvastatin in healthy male volunteers who receive metformin extended release alone, rosuvastatin alone, and both together in a 3 period repeatedly.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male volunteers, age 20 to 55 years.
2. The result of Body Mass Index(BMI) is not less than 19 kg/m2 , no more than 27 kg/m2
3. Subjects who have ability to comprehend the objectives, contents of study and property of study drug before participating in trial and have willingness to sign of informed consent in writing

Exclusion Criteria:

1. Presence of medical history or a concurrent disease that may interfere with treatment and safety assessment or completion of this clinical study, including clinically significant disorders in kidney, liver, cardiovascular system, respiratory system, endocrine system, or neuropsychiatric system.
2. Glomerular filtration rate is under 60ml/min which is calculated by serum creatinine value.
3. Liver enzyme (AST, ALT) level exceeds one and a half times more than maximum normal range.
4. Systolic blood pressure <90mmHg or Diastolic blood pressure < 60 mmHg, systolic blood pressure ≥ 140 mmHg or diastolic blood pressure ≥ 90 mmHg(Sitting blood pressure) during the screening procedure.

Ages: 20 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2013-01; Primary Completion 2013-03 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Metformin, Rosuvastatin Cmaxss | 0h(pre-dose), 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 9, 10, 12, 14, 24, 48 h of each period (total 16)
metformin, rosuvastatin AUC | 0h(pre-dose), 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 9, 10, 12, 14, 24, 48 h of each period (total 16)

SECONDARY OUTCOMES:
Metformin, Rosuvastatin tmaxss | 0h(pre-dose), 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 9, 10, 12, 14, 24, 48 h of each period (total 16)
Metformin, Rosuvastatin t1/2 | 0h(pre-dose), 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 9, 10, 12, 14, 24, 48 h of each period (total 16)
Metformin, Rosuvastatin C min,ss | 0h(pre-dose), 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 9, 10, 12, 14, 24, 48 h of each period (total 16)
Metformin, Rosuvastatin CL/Fss | 0h(pre-dose), 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 9, 10, 12, 14, 24, 48 h of each period (total 16)
Metformin, Rosuvastatin Vd/Fss | 0h(pre-dose), 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 9, 10, 12, 14, 24, 48 h of each period (total 16)

CONTACTS AND LOCATIONS:
Locations (1):
- Samgsung Seoul Hospital, Seoul, South Korea